CLINICAL TRIAL: NCT04704388
Title: Study Project Comparing the Sequelae of COVID-19 Infection in Patients Who Have and Have Not Received Ventilatory Support in Critical Care
Acronym: COMEBAC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: COMEBAC
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients hospitalized in intensive care units for SARS-CoV-2: patients hospitalized in intensive care units for SARS-CoV-2
- patients hospitalized outside intensive care units: patients hospitalized outside intensive care units

SUMMARY:
To assess the proportion of post-intensive care syndrome (PICS) of patients who received high flow humidified oxygen with FiO2 ≥50% for more than 48h and / or who received mechanical ventilation for more than 48h in a context of hospitalization in intensive care for COVID-19 pneumonia

ELIGIBILITY:
Inclusion Criteria:

-

Group 1: patients hospitalized in intensive care units for ARDS with SARS-CoV-2

* Major
* Admitted between March 1 and May 10, 2020 in one of the sectors of the Bicêtre hospital approved for critical care
* proven SARS-CoV-2 infection
* Treated by invasive mechanical ventilation or high flow humidified oxygen with FiO2 ≥50% for more than 48 hours.

Group 2: patients hospitalized outside intensive care units

* Major
* Admitted between March 1 and May 10, 2020 in an area of Bicêtre hospital having cared for patients infected with SARS-CoV-2 excluding critical care: pulmonology, internal medicine / orthopedics, infectious diseases, nephrology , acute geriatrics, neurology.

Exclusion Criteria:

* Patients having refused the post consultation at 3 month
* Without social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paitent admitted between March 1 and May 10, 2020 in Bicêtre hospital for an infection with SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
post-intensive care syndrome (PICS) | 3 month after hospitalisation
  To assess the proportion of post-intensive care syndrome (PICS) of patients who received high flow humidified oxygen with FiO2 ≥50% for more than 48h and / or who received mechanical ventilation for more than 48h in a context of hospitalization in intensive care for COVID-19 pneumonia.

SECONDARY OUTCOMES:
Evaluate the 3-month mortality of patients released alive from intensive care | 3 month after end of hospitalisation
  Number of patient deceased
Describe the overall state of health and the main organ sequelae of these patients | 3 month after hospitalisation
  Description of the data collected
functional respiratory sequelae | 3 month after hospitalisation
  Compare the functional respiratory sequelae of these patients to those who were hospitalized outside of critical care for COVID-19 pneumonia requiring lower oxygen support.

CONTACTS AND LOCATIONS:
Overall Officials: Tài PHAM, Principal Investigator — APHP
Locations (1):
- Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pham T, Morin L, Savale L, Colle R, Figueiredo S, Harrois A, Gasnier M, Lecoq AL, Meyrignac O, Noel N, Abdo A, Baudry E, Bellin MF, Beurnier A, Choucha W, Corruble E, Dortet L, Gosset E, Hardy-Leger I, Quinque M, Radiguer F, Sportouch S, Verny C, Wyplosz B, Zaidan M, Becquemont L, Montani D, Monnet X. Four- and sixteen-month clinical status of a cohort of patients following hospitalization for COVID-19. Respir Med Res. 2024 Nov;86:101099. doi: 10.1016/j.resmer.2024.101099. Epub 2024 Mar 4. PMID 38843604